# **Protocol Document**

Dose-response Effect of Dietary Nitrate on Muscle Function in Older Individuals

NCT03595774

June 3, 2019

# Dose-response effect of dietary nitrate on muscle function in older individuals

Principal Investigator: Andrew Coggan, Ph.D.

Associate Professor, Department of Kinesiology I.U. School of Health and Human Sciences

Sub-Investigators: Ranjani N. Moorthi, M.D.

Sharon Moe, M.D.

#### **Table of Contents:**

# **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/Exclusion Criteria
- 4.0 Enrollment/Randomization
- **5.0** Study Procedures
- **6.0** Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 7.0 Study Withdrawal/Discontinuation
- 8.0 Statistical Considerations
- 9.0 Privacy/Confidentiality Issues
- 10.0 Follow-up and Record Retention
- 11.0 References
- 12.0 Appendix

### 1.0 Background

By 2050, approximately 20% of the US population, or >80 million people, will be 65 y of age or older.¹ Unfortunately, aging is accompanied by a progressive reduction in the maximal strength, speed, and especially power of skeletal muscle. These age-related physiological changes often lead to functional limitations that are highly predictive of disability, institutionalization, and mortality in the elderly.²,³ Thus, any intervention that significantly enhances muscle contractile function could potentially improve the health, quality of life, and possibly even the longevity of older individuals.

Numerous factors undoubtedly account for the decline in muscle function described above, with age-related changes in the size, properties, and neural control of muscle likely all playing a role. Another important factor, however, may be a fall in NO bioavailability with aging. Although initially identified as a vasodilator, i.e., as "endothelium-derived relaxing factor", NO is in fact a key cellular signaling molecule with pleiotropic effects in many tissues. These include skeletal muscle, wherein among other effects NO helps modulate contractile function.<sup>5-9</sup> With aging, however, whole-body NO production decreases, as evidenced, e.g., by a progressive decline in the plasma concentrations of its downstream metabolites, NO<sub>2</sub> and NO<sub>3</sub>. <sup>10,11</sup> In skeletal muscle itself, there is a dramatic decrease in interstitial NO<sub>2</sub><sup>-</sup> and NO<sub>3</sub><sup>-</sup> concentrations, <sup>12</sup> as well as a decline in the activity of the neuronal form of NO synthase (nNOS, or NOS1),13,14 the primary isoenzyme within muscle responsible for the synthesis of NO from L-arginine, O2, and NADPH. These changes are accompanied by an age-related reduction in flow-mediated vasodilation, 15-18 perhaps the hallmark indicator of NO bioavailability. In turn, the latter (i.e., flow-mediated vasodilation) has been shown to correlate positively with muscular power and physical functioning in older men and women.<sup>19</sup> Taken together, these data suggest that decreased NO production may contribute to the ageassociated decline in muscle contractile properties and hence in functional capacity.

In this context, the physiological effects of dietary  $NO_3^-$  are of considerable interest. It is now recognized that, rather than being metabolically inert or, worse, a potential carcinogen,  $NO_3^-$  in the diet is a significant source of NO in the body (Fig. 1). In fact, this dietary pathway, which entails the reduction of  $NO_3^-$  to  $NO_2^-$  by facultative anaerobic bacteria in the mouth followed by further reduction of  $NO_2^-$  to NO by, e.g., deoxyhemoglobin, can account for as much as ~25% of basal whole-body NO production. This dietary pathway serves as an important "backup" system to the more well-known NOS pathway. This is likely to be especially true in skeletal muscle,

Figure 1. Enterosalivary pathway of NO production. From Ref. 22.



since unlike the NOS pathway the dietary pathway operates well at low pO<sub>2</sub> and is stimulated rather than inhibited by low pH,<sup>20-24</sup> conditions that regularly exist in muscle, both at rest and especially during contractile activity. Indeed, skeletal muscle has recently been shown to play a central role in whole-body NO<sub>3</sub>-/NO<sub>2</sub>-/NO metabolism.<sup>27,28</sup>

Based on the above, it is logical to hypothesize that <u>increased dietary</u> NO<sub>3</sub> intake <u>might enhance NO bioavailability in older men and women, leading to an improvement in the state of </u>

muscle function. Indeed, we have observed significant increases in muscle speed and power following dietary NO<sub>3</sub><sup>-</sup> intake in healthy younger subjects, <sup>29</sup> athletes, <sup>30</sup> and especially middle-aged heart failure patients. <sup>31</sup> (See Preliminary Data.) Along the same lines, Haider and Folland <sup>32</sup> and Whitfield et al. <sup>33</sup> have reported that dietary NO<sub>3</sub><sup>-</sup> intake enhances the rate of force development and peak force output of the quadriceps muscle of healthy young men during electrically-stimulated contractions. To date, however, no study has specifically examined the impact of dietary NO<sub>3</sub><sup>-</sup> on muscle contractile function in older persons. Furthermore, it cannot be automatically assumed that dietary NO<sub>3</sub><sup>-</sup> will be equally efficacious in older subjects. For example, in rodents the effects of dietary NO<sub>3</sub><sup>-</sup> are more prominent in fast- vs. slow-twitch muscle, <sup>34,35</sup> and some, <sup>36-39</sup> but not all, <sup>40-42</sup> studies of humans have found that aging results in a reduction in the percentage of fast-twitch muscle fibers. Alternatively and/or in addition, more rapid destruction of NO due to increased production of reactive oxygen species by aging muscle <sup>43</sup> could limit the beneficial effects of dietary NO<sub>3</sub><sup>-</sup> in older persons.

Even if the *efficacy* of a particular dose of NO<sub>3</sub><sup>-</sup> could be established in older subjects, this would not necessarily mean that it is the *optimal* dose. There is limited data in the literature regarding the dose-response relationship for dietary NO<sub>3</sub><sup>-</sup> for various outcomes, and only one study has examined the response to exercise over a wide range of doses.<sup>44</sup> These authors found that acute ingestion of either 8.4 or 16.8, but not 4.2, mmol of NO<sub>3</sub><sup>-</sup> improved performance equally during high intensity *aerobic* exercise in healthy young men. However, it is not known whether a similar plateau exists with respect to improvements in muscle contractile function, nor is it known whether aging influences this relationship. Such information is obviously critical to any attempt to pursue funding for larger (e.g., multicenter) trials evaluating dietary NO<sub>3</sub><sup>-</sup> as a potential treatment for reduced muscle function in older persons, especially since the incidence of negative side effects (e.g., GI distress) may increase at higher doses.

Our Preliminary Data (see below) suggest that older subjects may require a greater dose of NO<sub>3</sub><sup>-</sup> than younger individuals to yield a significant improvement in muscle speed and/or power.

#### Preliminary data

Using methods essentially identical to those to be employed in the proposed experiments (see below), we previously demonstrated that acute dietary  $NO_3^-$  intake increased maximal knee extensor speed (Vmax) and power (Pmax) in 12 healthy, younger men and women by  $11\pm5\%$  (P<0.05) and  $6\pm3\%$  (P<0.05), respectively.<sup>29</sup> We observed similar dietary  $NO_3^-$ -induced improvements in muscle speed and power in 13 athletes performing multi-joint, multi-muscle, i.e., sprint cycling, exercise.<sup>30</sup> Lastly, we found even greater increases in Vmax and Pmax (of  $12\pm5\%$ , P=0.09, and  $13\pm4\%$ , P<0.05, y) in nine middle-aged patients with systolic heart failure (HF).<sup>31</sup>

Using the same methods, we have also recently determined the effects of dietary  $NO_3^-$  in six healthy men and women 64-79 y of age. As shown in Table 1, plasma  $NO_3^-$  and  $NO_2^-$  and breath NO increased (P<0.05) by  $1309\pm188\%$ ,  $268\pm91\%$ , and  $142\pm19\%$ , respectively, by 2 h after ingestion, and all three remained elevated for the remainder of the experiment. These findings are consistent with our previous research.<sup>29-31</sup> This increase in NO bioavailability resulted in a 9±5% increase in maximal muscle speed, i.e., Vmax (Fig. 2, *left panel*), with five out of the six subjects demonstrating an improvement. This increase, however, was not statistically significant (i.e., P=0.13), and maximal muscle power, i.e., Pmax, improved on average by only  $2\pm3\%$ 

<u>Table 1. Changes in plasma  $NO_3^-$  and  $NO_2^-$  and breath NO in response to dietary  $NO_3^-$  intake in older study participant.</u>

| | Trial | <u>Pre</u> | 1 h | <u>2 h</u> | 10 min post |
|---|---|---|---|---|---|
| | <u>ITIGI</u> | <u>11C</u> | <u> 1 11</u> | <u>2 11</u> | <u>exercise</u> |
| Plasma NO₃⁻ | Placebo | 26±4 | 24±3 | 24±3 | 22±4 |
| (µmol/L) | Nitrate | 31±7 | 285±27* | 295±27* | 282±33* |
| Plasma NO <sub>2</sub> - | Placebo | $0.21 \pm 0.03$ | $0.26 \pm 0.06$ | $0.26 \pm 0.06$ | $0.20\pm0.03$ |
| (µmol/L) | Nitrate | $0.27 \pm 0.04$ | $0.43 \pm 0.13$ | 0.49±0.06* | 0.56±0.10* |
| <b>Breath NO</b> | Placebo | 23±5 | 26±4 | 27±4 | 23±5 |
| (ppb) | Nitrate | 27±4 | 49±7* | 38±4* | 52±10* |

Values are mean  $\pm$  S.E. for n=7. \*Nitrate trial significantly higher than Placebo trial at same time point (P<0.05).

(P=0.47) (Fig. 2, *center panel*). This is only 1/3<sup>rd</sup> as much as we previously found in younger Figure 2. Responses of Vmax (left panel) and Pmax (center and right panels) to dietary NO<sub>3</sub> in older subjects.



men and women.  $^{29,30}$  Closer examination of the data suggested that this diminished effect was due to an inadequate dose of  $NO_3^-$ , as there was a significant positive relationship between  $NO_3^-$  intake relative to body mass and the relative improvement in Pmax (Fig. 2, *right panel*). These preliminary results therefore suggest that older individuals remain responsive to  $NO_3^-$ , but that a higher dose may be required to elicit improvements in muscle contractile function.

#### 2.0 Rationale and Specific Aims

In light of the above, we will use a double-blind, placebo-controlled, crossover design to address the following Specific Aim:

#### Specific Aim #1:

To determine the dose-response relationship between acute dietary  $NO_3^-$  supplementation and muscle contractile function in healthy, older (i.e., 65-79 y old) men and women.

#### 3.0 Inclusion/Exclusion Criteria

#### Inclusion:

- Men and women age 65-79
- In good health, as determined by the physician's review of history, physical examination, resting EKG, and routine blood tests

#### Exclusion:

- Men and women <65 or >79 years of age
- Unable to provide informed consent
- Currently pregnant or lactating

- Current smokers
- Significant orthopedic limitations or other contraindications to strenuous exercise
- Those taking phosphodiesterase inhibitors (e.g., Viagra)
- Those taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy
- History of major metabolic disease (e.g., type I and type II diabetes, thyroid disorders),
   history of neuromuscular disease (e.g., cervical spondylotic radiculomyelpathy, lumbar

#### Figure 3. Study design.

spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies), cardiovascular disease (e.g., > stage II hypertension, heart failure, myocardial infarction/ischemia, significant myocardial or pericardial diseases (e.g. amyloidosis, constriction), moderate or severe valvular disease, renal disease, liver disease, or anemia

Twenty study participants will be enrolled.

#### 4.0 Enrollment/Randomization

Subjects will be recruited from the community through approved methods including flyers, emails from the Indiana Clinical and Translational Sciences Institute (All IN for Health), and being included in the searchable "All IN for Health" clinical trials database . When potential study subjects contact the study team expressing an interest in the study they will be given additional information regarding the study procedures, requirements, and risks. If they are still interested the study team will complete a brief phone screening to see if they qualify for an in-person screening visit. As previously approved by amendment, potential subjects will be asked if they are part of the IU Health medical system and if so, do they give verbal permission for their records to be reviewed for possible exclusions to participation. If they are not part of the IU Health system or do not give permission, they will still be able to participate in a screening visit if it appears they meet other pre-screening criteria. If it appears they are eligible for a screening visit, they will be scheduled and a consent form will be mailed / emailed to them ahead of the screening visit for review. After the study participant has had several days to review the consent form, a study team member will call to answer any questions the participant may have regarding the consent form. When the subject arrives for the screening visit a member of the research team will thoroughly review the consent with the study participant and answer questions. Study participants will be given as much time as they wish to consider participation before signing the consent form. If the study participant agrees to move forward with the screening visit, the consent will be signed by the study participant and the person who reviewed the consent and obtained the participant's signature. A copy of the signed consent form will be provided. Both the participants and the investigators will be blinded to the order of treatment, which will be randomized using randomization.com.

#### 5.0 Study Procedures

#### Study Design

Each subject will be studied using a double-blind, placebo-controlled, crossover design. Figure 3 illustrates the flow through the study for an individual participant.



#### Study Procedures

Participants will be asked to fast for 12 hours prior to each study day.

**On Study Day 1** (Pre-test), all study participants will complete a screening / phenotyping examination. The participant will undergo a complete history, physical exam, resting EKG and phlebotomy for screening and phenotyping laboratories (complete blood count, liver and kidney function tests, electrolytes, fasting glucose and insulin). They will also practice the entire isokinetic dynamometer exercise test.

To minimize variation in baseline  $NO_3^-/NO_2^-/NO$  levels, participants will be instructed to consume their normal diet (aside from the BRJ supplement) throughout the study. Participants will, however, be asked to avoid consumption of high  $NO_3^-$  foods (e.g., beets, spinach, collard greens) the evening prior to testing. This approach is justified based on the short half-life of  $NO_3^-$  in plasma (i.e.,  $\sim 8$  h) as well as previous research demonstrating that even a chronic increase in dietary  $NO_3^-$  intake up to 2.5 mmol/d (i.e.,  $\sim 3x$  normal dietary  $NO_3^-$  intake in the US) has no significant influence. For Participants will be asked to refrain from chewing gum, alcohol, and caffeine-containing food/drinks for 24 h prior to each remaining visit. Participants will also be instructed to refrain from use of an antibacterial mouthwash throughout the study, since this would limit conversion of  $NO_3^-$  to  $NO_2^-$  by bacteria in the oral cavity. Participants will be asked to fast for 12 h prior to each remaining study visit.

On Study Day 2, participants will undergo phlebotomy for plasma NO<sub>3</sub><sup>-</sup> and NO<sub>2</sub><sup>-</sup> measurement, and have their breath NO level determined. (Breath NO will be measured as a biomarker of increases in whole-body NO production in response to dietary NO<sub>3</sub>- intake.<sup>52,53</sup>) The subject will then ingest 3.3 mL/kg of a commercial concentrated beetroot juice (BRJ) supplement (Beet It Sport<sup>®</sup>, James White Drinks, Ipswich, UK) either: 1) essentially devoid of NO<sub>3</sub><sup>-</sup> (placebo); 2) containing (as determined by previous direct measurement) 91 µmol/mL NO<sub>3</sub>- (thus total dose = 300 µmol/kg, or 21 mmol in a 70 kg subject); or 3) an equal mixture of the placebo and NO<sub>3</sub>containing BRJ products. The placebo, which is prepared the company by extracting NO<sub>3</sub>- from BRJ using an ion exchange resin, is indistinguishable in packaging, color, taste, texture, and smell from the standard product, and does not alter plasma NO<sub>3</sub><sup>-</sup>/NO<sub>2</sub><sup>-</sup> or breath NO concentrations or the physiological responses to exercise.<sup>29-31</sup> Additional blood and breath samples will be obtained 1 and 2 h later, as well as blood pressure and heart rate, afterwhich time the subject will have the Vmax and Pmax of the knee extensor muscles of their dominant leg determined via isokinetic dynamometry (see below). The timing of all measurements has been chosen to correspond to peak plasma NO<sub>3</sub>-/NO<sub>2</sub>- concentrations and breath NO levels, which reach a maximum 2-3 h after ingestion.<sup>29-31</sup>

**On Study Days 3 and 4**, participants will be asked to return to undergo the same studies as described above for Study Day 2.

Study Methods

Measurement of  $NO_3^-$  in each batch of BRJ w/ or w/o  $NO_3^-$ : The  $NO_3^-$  content of each batch of BRJ w/ or w/o  $NO_3^-$  will be determined using high performance liquid chromatography (HPLC) (ENO-30, Eicom USA, San Diego, CA).

Measurement of plasma  $NO_3^-$ ,  $NO_2^-$ , and breath NO: Venous blood samples will be obtained prior to consumption of BRJ w/ or w/o  $NO_3^-$  and every hour thereafter for 3 hours, plasma rapidly separated by centrifugation, and frozen at -80° C until subsequently analyzed for  $NO_3^-$  and  $NO_2^-$  concentration using HPLC as described above. Breath NO levels will be measured at the same time points using a portable electrochemical analyzer (NIOX VERO, Circassia Pharmaceuticals, Chicago, IL).

Measurement of skeletal muscle contractile function: A Biodex 4 system will be used to measure each subject's muscle contractile properties as previously described.<sup>29-31</sup> Briefly, subjects will perform maximal knee extensions with their dominant leg at angular velocities of 0, 1.57, 3.14, 4.71, and 6.28 rad/s. (Not all older individuals may be able to achieve the highest velocity – if not, the highest measured angular velocity and associated torque will be used in all subsequent calculations.) The subject will perform 3-4 knee extensions at each velocity, with 2 min of rest allowed between each set of contractions. To eliminate artifacts, data will be "windowed" to isolate the isokinetic phase and smoothed using a 9 point weighted moving average filter. The highest torque generated at each velocity will be used to calculate peak power at that velocity, after which the resulting power-velocity curve will be fit to a polynomial function to determine the subject's maximal knee extensor velocity (Vmax) and corresponding power (Pmax). Subsequently, the subject will perform an "all out" 50 contraction fatigue test (at 3.14 rad/s) to determine whether dietary NO<sub>3</sub><sup>-</sup> influences fatigue resistance (i.e., increases average power) during repetitive, maximal activation. Finally, recovery of muscle function will be quantified by measuring restoration of torque during knee extensions performed periodically over the next 10 min.

# **Risks**

Likely: The insertion of an intravenous tube for blood drawing is associated with a small amount of discomfort. The subjects are likely to notice reddish urine or stools after drinking beetroot juice or control. This is normal and not harmful.

Less Likely: The insertion of an intravenous tube for blood drawing is associated with a small risk of bleeding or infection. After the EKG, some people may experience a skin rash but this usually goes away without treatment.

Rare: The risk of arrhythmia and heart attack are rare and the risk of death during exercise testing is extremely rare. The risk of heart attack is <0.1% in all patients undergoing exercise testing (and should be lower in these subjects since they have no coronary artery disease). The risk of death is reported as less than 2/10,000 tests or <0.02%.

#### Mitigation of Risks

Blood draw: Only trained staff will place IVs and collect blood samples

EKG: trained nurses will prepare the skin for the EKG and place the electrodes.

Exercise test: Every effort to minimize these rare risks by observing and monitoring during testing. Emergency equipment and trained personnel are available to deal with any emergency.

# 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

The following standard definitions will be used for this study:

Adverse event (AE): Any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.

Serious Adverse Event (SAE): Any AE that results is place the participant at immediate risk of death from the event as it occurred, or results in inpatient hospitalization, prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital abnormalities or birth defects, or death.

Unanticipated problem: As Defined by DHHS 45 CFR part 46, any incident, experience, or outcome that meets all of the following criteria: 1) is unexpected, in terms of nature, severity, or frequency, given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the study population; 2) is related or possibly related to participation in the research (in this guidance document, possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and 3) suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

AEs will be graded according to the following scale:

- <u>Mild</u>: An experience that is transient, and requires no special treatment or intervention. The experience does not generally interfere with usual daily activities. This includes transient laboratory test alterations.
- <u>Moderate</u>: An experience that is alleviated with simple therapeutic treatments. The
  experience impacts usual daily activities. Includes laboratory test alterations indicating
  injury, but without long-term risk.
- <u>Severe</u>: An experience that requires therapeutic intervention. The experience interrupts usual daily activities. If hospitalization (or prolongation of hospitalization) is required for treatment it becomes an SAE.

Attribution of AEs and SAEs will be categorized as:

- <u>Not related</u>: The AE is clearly not related to the study procedures (i.e., another cause of the event is most plausible and/or a clinically plausible temporal sequence is inconsistent with the onset of the event).
- <u>Possibly related</u>: An event that follows a reasonable temporal sequence from the initiation
  of study procedures, but that could readily have been produced by a number of other
  factors.
- Related: The AE is clearly related to the study procedures.

Reporting of AEs, SAEs, and unanticipated problems will follow the guidelines of the IU Standard Operating Procedure for Reporting Unanticipated Problems and Noncompliance. Specifically, the following events will be reported promptly (i.e., within five business days) to the IRB:

- AEs (including SAEs) that are assessed by the PI or coinvestigators as (1) unexpected, (2) related or possibly related to participation, AND (3) suggests that the research places subject(s) or others at greater risk of harm than was previously known;
- *Major protocol deviations* that may, in the opinion of the PI, (1) impact subject safety, (2) affect the integrity of the data, OR (3) affect study participant' willingness to participate in the study;
- Noncompliance, which includes any action or activity associated with the conduct or oversight of the research that fails to comply with federal or state regulations, institutional policies governing human study participant research, or the requirements or determinations of the IRB.

Unanticipated problems that do not meet the criteria for prompt reporting will be reported at time of protocol renewal to ensure the IRB has a full understanding of the conduct of the research

#### **Study Withdrawal/Discontinuation**

A participant may withdrawal from the study at any time verbally or by providing this request in writing as described in the informed consent document. As outlined in the consent document, if the participant/patient wishes to withdraw consent, the PI will:

- no longer use and take reasonable steps to destroy all blood/tissue samples and information
- not take back any research / analyses already completed

#### 7.0 Statistical Considerations

Statistical analyses: Normality of data distribution will first be tested using the D'Agostino-Pearson omnibus test. Analysis of individual endpoints will then be conducted using a mixed model analysis of variance (ANOVA) approach, with dose, trial number, and sequence as fixed effects and subject as a random effect to account for repeated measurements. As a preliminary analysis, carryover will be evaluated by testing the effect of sequence, i.e. does the effect of dose depend on trial. Assuming a sufficient washout period, i.e., no carryover effect, analysis of dose will proceed using all trials. Dose effects will be determined from ANOVA model results. A P value of <0.05 will be considered significant.

Calculation of sample size/power analyses. Our proposed sample size (i.e., n=20) for this pilot, proof-of-concept study has been chosen primarily based on budgetary considerations and the 1 y duration of the project. G\*Power® version 3.1.9.4<sup>59</sup> was used to determine the sample size required to provide a power (i.e., 1-B) of 0.90 assuming an effect size (i.e., Cohen's d) of 1.5. This effect size is based on the n=7 healthy older subjects that we have studied to date and is roughly the same as that we have previously observed for the effects of dietary  $NO_3^-$  on muscle contractile function in younger subjects.<sup>29,30</sup> These calculations demonstrated that with  $\alpha=0.05$ , n=15 would be sufficient to provide the chosen power. The power that a sample size of n=15 would provide to detect other effect sizes is shown in Figure 4. Based on these calculations, we will enroll 20 subjects to allow for subject drop-out.

Potential limitations and alternatives considered: A possible limitation of the proposed study is the lack of direct demonstration that dietary NO<sub>3</sub><sup>-</sup> results in an increase in NO specifically within muscle. This is because 1) the biological half-life of NO is extremely short (i.e., seconds), precluding measurement of its concentration in human tissue samples, and 2) existing stable isotopic methods only measure the rate of NO production via the NOS pathway, and not the enterosalivary pathway. We will, however, measure changes in plasma NO<sub>3</sub><sup>-</sup>/NO<sub>2</sub><sup>-</sup> and breath NO (a biomarker of whole-body NO bioavailability) levels in response to dietary NO<sub>3</sub><sup>-</sup>. We therefore do not consider the absence of direct measurements of plasma or muscle NO a significant limitation.



A more significant limitation of the proposed study is that, due to budgetary and time constraints, we will be evaluating only two doses of NO<sub>3</sub>. We will therefore be unable to identify the truly optimal dose (which could fall inbetween the two doses to be tested, or higher than the highest dose). As stated previously, however, there is very limited data in the literature regarding the dose-response relationship of dietary NO<sub>3</sub>, especially with respect to changes in exercise performance. Thus, despite this limitation the information to

be gained from this study will represent a significant advance, and in fact is a necessary first step towards the design of larger (e.g., multicenter) studies.

By focusing specifically on changes in muscle contractile properties, we will not be able to determine whether dietary  $NO_3^-$  supplementation reduces the  $O_2$  cost of exercise in older subjects. We will also not be measuring the effect of acute and/or chronic dietary  $NO_3^-$  intake on muscle blood flow, or on muscle energetics or aerobic exercise performance. We will also not be testing whether dietary  $NO_3^-$  intake improves insulin sensitivity. Several recent studies, however, have reported that dietary  $NO_3^-$  (or  $NO_2^-$ ) does not significantly improve aerobic exercise function in older men and women.  $^{60-63}$  (Despite increasing muscle contractile function.  $^{63}$ ) Similarly, several other recent studies have demonstrated that, contrary to the results of *in vitro* experiments,  $^{64}$  dietary  $NO_3^-$  does not enhance insulin sensitivity in older humans.  $^{65-67}$  We therefore believe that we are well-justified in focusing on changes in muscle contractile properties, especially in light of the important role that reductions in muscle function play in the aging process.

Because our focus is muscle contractile function, we considered using percutaneous electrical nerve stimulation rather than voluntary exercise. However, this approach inverts the normal orderly recruitment of motor units, preferentially depolarizing larger alpha motor neurons innervating type II muscle fibers.  $^{68}$  Thus, while potentially magnifying the effects of dietary  $NO_3$  on muscle speed and power it would significantly diminish the external validity of our findings.

Although the proposed study will provide important new information regarding the effect of NO<sub>3</sub><sup>-</sup> dose on muscle contractile function in older individuals, it will not address the mechanism(s) responsible for any improvements that may be observed. While clearly relevant, answering such questions are beyond the scope of the present investigation.

Finally, we note that historically there have been concerns that increased NO<sub>3</sub><sup>-</sup> intake may lead to formation of carcinogenic nitrosamines.<sup>69</sup> However, the Joint FAO/WHO Expert Committee on Food Additives has concluded that "Overall, the epidemiological studies showed no consistently

increased risk for cancer with increasing consumption of  $NO_3^-$ ." Furthermore, diets high in vegetables, such as the DASH diet widely recommended to hypertensive patients, routinely exceed the WHO acceptable daily intake of  $NO_3^-$  by >5-fold. In contrast, the amount of dietary  $NO_3^-$  shown to improve exercise tolerance in previous studies is only slightly above the WHO limit. Nonetheless, the safety and efficacy of increased dietary  $NO_3^-$  would need to be established in follow-up large-scale, longer-term studies before BRJ or other  $NO_3^-$ -rich foods or could be widely recommended to older individuals.

## 8.0 Privacy/Confidentiality Issues

All study activities will be performed within areas respective of the participants' right to privacy.

Although there can be no absolute guarantee of confidentiality, every practical precaution will be taken.

Each study participant will be assigned a unique ID. Samples and information will be de-identified using this unique ID.

#### 9.0 Follow-up and Record Retention

Study recruitment will be ongoing. The duration of the entire study is expected to be 12 months.

Any remaining blood samples will be de-identified and discarded. The de-identified data will be retained on computer files indefinitely. Hard copy study documents will be kept in a locked, file cabinet in a locked room. Electronic study information will be stored on a specified, password-protected network that is backed up daily. Only the study team and the relevant personnel will have access. Files will be kept on site until 2 years after study completion, and then sent to a secure archiving facility. Files will be kept for 7 years after study completion per state law requirements.

#### 10.0 References

- 1. Projections of the Population by Selected Age Groups and Sex for the United States: 2010 to 2050 (NP2008-T2) Population Division, U.S. Census Bureau (2008).
- 2. Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol 1994;49:M85–M94.
- 3. Kokkinos P, Myers J. Exercise and physical activity: clinical outcomes and applications. Circulation 2010;122:1637–1648.
- 4. Reid KF, Fielding RA. Skeletal muscle power: A critical determinant of physical functioning in older adults. Exerc Sports Sci Rev 2012:40:4-40. PMCID:PMC3245773.
- 5. Kaminski HJ, Andrade FH. Nitric oxide: biologic effects on muscle and role in muscle diseases. Neuromuscular Disord 2001;11:517-524.
- 6. Maréchal G, Gaily P. Effects of nitric oxide on the contraction of skeletal muscle. Cell Mol Life Sci 1999;55:1088-1102.
- 7. Stamler JS, Meissner G. Physiology of nitric oxide in skeletal muscle. Physiol Rev 2001;81:209-237.
- 8. Suhr S, Gehlert S, Gau M, Bloch W. Skeletal muscle function during exercise fine-tuning of diverse subsystems by nitric oxide. Int J Mol Sci 2013;14:7109-7139. PMCID: PMC3645679.

- 9. Lamb GD, Westerblad H. Acute effects of reactive oxygen and nitrogen species on the contractile function of skeletal muscle. J Physiol 2011;589:2119-2127. PMCID: PMC3098691
- 10. Di Massimo C, Lo Presti R, Corbacelli C, Pompei A, Scarpelli P, De Amicis D, Caimi G, Tozzi Ciancarelli MG. Impairment of plasma nitric oxide availability in senescent healthy individuals: Apparent involvement of extracellular superoxide dismutase activity. Clin Hemorheol Microcirc 2006;35:231–237.
- 11. Di Massimo C, Scarpelli P, Di Lorenzo N, Caimi G, di Orio F, Ciancarelli MG. Impaired plasma nitric oxide availability and extracellular superoxide dismutase activity in healthy humans with advancing age. Life Sci 2006;78:1163-1167.
- 12. Nyberg M, Blackwell JR, Damsgaard R, Jones AM, Hellsten Y, Mortensen SP. Lifelong physical activity prevents an age-related reduction in arterial and skeletal muscle nitric oxide bioavailability in humans. J Physiol 2012;590:5361-5370. PMCID: PMC3515824.
- 13. Richmonds CR, Boonyapisit K, Kusner LL, Kaminski HJ. Nitric oxide synthase in aging rat skeletal muscle. Mech Aging Dev 1999;109:177-189.
- 14. Song W, Kwak H-B, Kim J-H, Lawler JM. Exercise training modulates the nitric oxide synthase profile in skeletal muscle from old rats. J Gerontol A Biol Sci Med Sci 2009;64A:540-549. PMCID: PMC2800810.
- 15. Scrage WE, Eisenach JH, Joyner MJ. Aging reduces nitric oxide- and prostaglandin-mediated vasodilation in exercise humans. J Physiol 2007;579:227-236. PMCID: PMC2075375.
- 16. Proctor DN, Parker BA. Vasodilation and vascular control in contracting muscle of the aging human. Microcirculation 2006;13:315-327.
- 17. Behnke BJ, Delp MD. Aging blunts the dynamics of vasodilation in isolated skeletal muscle resistance vessels. J Appl Physiol 2010;108:14-20. PMCID:PMC2885069.
- 18. Hirai DM, Copp SW, Holdsworth CT, Ferguson SK, Musch TI, Poole DC. Effects of neuronal nitric oxide synthase inhibition on microvascular and contractile function in skeletal muscle of aged rats. Am J Physiol Heart Circ Physiol 2012;303:H1076-1084. PMCID:PMC3469646.
- 19. Heffernan KS, Chalé A, Hau C, Cloutier GJ, Phillips EM, Warner P, Nickerson H, Reid KF, Kuvin JT, Fielding RA. Systemic vascular function is associated with muscular power in older adults. J Aging Res 2012:2012:386387. Published online 2012 August 26. doi: 10.1155/2012/386387. PMCID:PMC3433136.
- 20. Lundberg JO, Weitzberg E, Gladwin MT. The nitrate—nitrite—nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov 2008;7:156-167.
- 21. Lundberg JO, Weitzbefg E. NO generation from inorganic nitrate and nitrite: Role in physiology, nutrition, and therapeutics. Arch Pharm Res 2009;32:1119-1126.
- 22. Lundberg JO, Weitzberg E. NO-synthase independent NO generation in mammals. Biochem Biophys Res Commun 2010;396:39-45.
- 23. Gilchrist M, Winyard PG, Benjamin N. Dietary nitrate--good or bad? Nitric Oxide 2010;22:104-109.
- 24. Machha A, Schecter AN. Dietary nitrite and nitrate:a review of potential mechanisms of cardiovascular benefits. Eur J Nutr 2011;50:293-303. PMCID:PMC3489477.
- 25. Wagner DA, Schultz DS, Deen WM, Young VR, Tannenbaum SR. Metabolic fate of an oral dose of <sup>15</sup>N-labeled nitrate in humans: Effect of diet supplementation with ascorbic acid. Cancer Res 1983;43:1921-1925.
- 26. Siervo M, Stephan BCM, Feelisch M, Bluck LJC. Measurement of in vivo nitric oxide synthesis in humans using stable isotopic methods: a systematic review. Free Radical Bio Med 2011;51:795-804.
- 27. Piknova B, Park JW, Swanson KM, Dey S, Noguchi CT, Schechter AN. Skeletal muscle as an endogenous nitrate reservoir. Nitric Oxide 2015;47:10-16. PMCID: PMC4439352.

- 28. Piknova B, Park JW, Kwan JLK, Schechter AN. Nitrate as a source of nitrite and nitric oxide during exercise hyperemia in rat skeletal muscle. Nitric Oxide 2016;55-56:54-61. PMCID: PMC4860042.
- 29. Coggan AR, Leibowitz JL, Kadkhodayan A, Thomas DT, Ramamurthy S, Anderson Spearie C, Waller S, Farmer M, Peterson LR. Effect of acute dietary nitrate intake on knee extensor speed and power in healthy men and women. Nitric Oxide 2015;48:16-21. PMCID: PMC4362985.
- 30. Rimer EG, Peterson LR, Coggan AR, Martin JC. Acute dietary nitrate supplementation increases maximal cycling power in athletes. Int J Sports Physiol Perf 2016;11:715-720. PMCID: 4889556.
- 31. Coggan AR, Leibowitz JL, Anderson Spearie C, Kadkhodayan A, Thomas DP, Ramamurthy S, Mahmood K, Park S, Waller S, Farmer M, Peterson LR. Acute dietary nitrate intake improves muscle contractile function in patients with heart failure: a double-blind, placebo-controlled, randomized trial. Circ Heart Fail 2015;8:914-920. PMCID: PMC4573847.
- 32. Haider G, Folland JP. Nitrate supplementation enhances the contractile properties of human skeletal muscle. Med Sci Sports Exerc 2014; 46:2234-2243.
- 33. Whitfield J, Gamu D, Heigenhauser GJF, Van Loon LJC, Spriet LL, Tupling AR, Holloway GP. Beetroot juice increases human muscle force without changing Ca<sup>2+</sup>-handling proteins in humans. Med Sci Sports Exerc. 2017; 49:2016-2024.
- 34. Ferguson AK, Hirai DM, Copp SW, Holdsworth CT, Allen JD, Jones AM, Musch TI, Poole DC. Impact of dietary nitrate supplementation via beetroot juice on exercising muscle vascular control in rats. J Physiol 2013;591:547-555. PMCID: PMC3577528.
- 35. Hernández A, Schiffer TA, Ivarsson N, Cheng AJ, Bruton JD, Lundberg JO, Weitzberg E, Westerblad H. Dietary nitrate increases tetanic [Ca<sup>2+</sup>]<sub>I</sub> and contractile force in mouse fast-twitch muscle. J Physiol 2012;590:3575-3583. PMCID: PMC3547271.
- 36. Larsson L, Grimby G, Karlsson J. Muscle strength and speed of movement in relation to age and muscle morphology. J Appl Physiol 1979;46:451-456.
- 37. Lexell J. Human aging, muscle mass, and fiber type composition. J Gerontol A Biol Sci Med Sci 1995;50A:11-16.
- 38. Lee WS, Cheung WH, Qin L, Tang N, Leung KS. Age-associated decrease of type IIA/B human skeletal muscle fibers. Clin Orthop Relat Res 2006;450:231-237.
- 39. Marzani B, Felzani G, Bellomo RG, Vecchiet J, Marzatico F. Human skeletal muscle aging: ROS-mediated alterations in rectus abdominis and vastus lateralis muscles. Exp Gerontol 2005;40:959-965.
- 40. Coggan AR, Spina RJ, Rogers MA, King DS, Brown M, Nemeth PM, Holloszy JO. Histochemical and enzymatic comparison of the gastrocnemius muscle of young and elderly men and women. J Geront 1992;47:B71-B76.
- 41. Frontera WR, Reid KF, Phillips EM, Krivickas LS, Hughes VA, Roubenoff R, Fielding RA. Muscle fiber size and function in elderly humans: a longitudinal study. J Appl Physiol 2008;105:637-642. PMCID: PMC2519941.
- 42. Verdijk LB, Dirks ML, Snijders T, Prompers JJ, Beelen M, Jonkers RA, Thijssen DH, Hopman MT, Van Loon LJ. Reduced satellite cell numbers with spinal cord injury and aging in humans. Med Sci Sports Exerc 2012;44:2322-2330.
- 43. Doria E, Buonocore D, Focarelli A, Marzatico F. Relationship between human aging muscle and oxidative system pathway. Oxid Med Cell Longev 2012;2012:803257. Doi: 10.1155/2012/830257. Epub 2012 May 17.
- 44. Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and dose-response relationships. J Appl Physiol 2013;115:325-336.

- 45. Jones AM, Bailey SJ, Vanhatalo A. Dietary nitrate supplementation and exercise performance. Sports Med 2014;44:S35-S45.
- 46. Stweart AL, Mills KM, King AC, Haskell WL, Gillis D, and Ritter PL. CHAMPS Physical Activity Questionnaire for Older Adults: outcomes for interventions. Med Sci Sports Exerc 2001; 33:1126-1141.
- 47. Webb DJ, Freestone S, Allen MJ, Muirhead GJ. Sildenafil citrate and blood-pressure-lowering drugs: results of drug interaction studies with an organic nitrate and a calcium antagonist. Am J Cardiol 1999; 83:21C-28C.
- 48. Lundberg JO, Weitzberg E, Lundberg JM, Alving K. Intragastic nitric oxide production in humans: measurements in expelled air. Gut 1994; 35:1543-1546.
- 49. Obach RS, Huynh P, Allen MC, Beedham C. Human liver aldehyde oxidase: inhibition by 239 drugs. J Clin Pharmacol 2004;44:7-19.
- 50. Levey AS, Stevens LA, Schmid CH, et al. A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009;150:604-612.
- 51. Levey AS, Stevens LA. Estimating GFR using the CKD Epidemiology Collaboration (CKD-EPI) creatinine equation: more accurate GFR estimates, lower CKD prevalence estimates, and better risk predictions. Am J Kidney Dis. 2010;55:622-627.
- 52. Olin AC, Aldenbratt A, Ekman A, Ljungkvist G, Jungersten L, Alving K, Torén K. Increased nitric oxide in exhaled air after intake of a nitrate-rich meal. Resp Med 2001;95:153-158.
- 53. Vints AM, Oostveen E, Eeckhaut G, Smolders M, De Backer WA. Time-dependent effect of nitrate-rich meals on exhaled nitric oxide in healthy subjects. Chest 2005;128;2465-70.
- 54. Griesenbeck JS, Steck MD, Huber JC Jr, Sharkey JR, Rene AA, Brender JD. Development of estimates of dietary nitrates, nitrites, and nitrosamines for use with the Short Willet Food Frequency Questionnaire. Nutr J. 2009;8:16. doi:10.1186/1475-2891-8-16. PMCID: PMC2669451.
- 55. Kapil V, Milsom AB, Okorie M, Maleki-Toyserkani S, Akram F, Rehman F, Arghandawi S, Pearl V, Benjamin N, Loukogeorakis S, Macallister R, Hobbs AJ, Webb AJ, Ahluwalia A. Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO. Hypertension 2010; 56:274-281.
- 56. Miller GD, Marsh AP, Dove RW, Beavers D, Presley T, Helms C, Bechtold E, King BS, Kim-Shapiro D. Plasma nitrate and nitrite are increased by a high-nitrate supplement but not by high-nitrate foods in older adults. Nutr Res 2012;32:160-168. PMCID: PMC3319660.
- 57. Govoni M, Jansson EA, Weitzberg E, Lundberg JO. The increase in plasma nitrite after a dietary nitrate load is markedly attenuated by an antibacterial mouthwash. Nitric Oxide 2008;19:333-337.
- 58. American Thoracic Society/European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med 2005;171:912–930.
- 59. Faul F, Erdfelder E, Lang AG, Buchner A. G\*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007;39:175–191. doi: 10.3758/BF03193146.
- 60. Kelly J, Fulford J, Vanhatalo A, Blackwell JR, French O, Bailey SJ, Gilchrist M, Winyard PG, Jones AM. Effects of short-term dietary nitrate supplementation on blood pressure, O₂ uptake kinetics, and muscle and cognitive function in older adults. Am J Physiol Regul Integr Comp Physiol 2013;304:R73−R83.
- 61. Siervo M, Oggioni C, Jakovljevic DG, Trenell M, Mathers JC Houghton D, Celis-Morales C, Ashor AW, Ruddock A, Ranchordas M, Klonizakis M, Williams EA. Dietary nitrate does not

- affect physical activity or outcomes in healthy older adults in a randomized, cross-over trial. Nutr Res 2016; 36:1361-1369.
- 62. Shaltout HA, Eggebeen J, Marsh AP, Brubaker PH, Laurienti, PJ, Burdette JH, Basu S, Morgan A. Dos Santos PC, Norris JL, Morgan TM, Miller GD, Rejeski WJ, Hawfield AT, Diz DI, Becton JT, Kim-Shapiro DB, Kitzman DW. Effects of supervised exercise and dietary nitrate in older adults with controlled hypertension and/or heart failure with preserved ejection fraction. Nitric Oxide 2017; http://dx.doi.org/10.1016/j.niox.2017.05.005.
- 63. Justice JN, Johnson LC, DeVan AE, Cruickshank-Quinn C, Reisdorph N, Bassett CJ, Evans TD, Brooks FA, Bryan NS, Chonchol MB, Giordano T, McQueen MB, Seals DR. Improved motor and cognitive performance with sodium nitrite supplementation is related to small metabolite signatures: a pilot trial in middle-aged and older adults. Aging 2015; 7:1004-1021.
- 64. Deshmukh As, Long YS, de Castro Barbosa E, Karlsson HKR, Glund S, Zavadoski WJ, Gibbs Em, Koistinen HA, Wallberg-Henricksson H, Zierath JR. Nitric oxide increases cyclic GMP levels, AMP-activated protein kinase (AMPK)a1-specific activity and glucose transport in human skeletal muscle. Diabetolog 2010;53:1142-1150. PMCID: PMC2860569.
- 65. Gilchrist M, Winyard PG, Aizawa K, Anning C, Shore A, Benjamin N. Effect of dietary nitrate on blood pressure, endothelial function, and insulin sensitivity in type 2 diabetes. Free Radic Bio Med 2013; 60:89-97.
- 66. Cermak NM, Hansen D, Kouw IW, van Dikk JW, Blackwell JR, Jones AM, Gibala MJ, va Loon LJ. A single dose of sodium nitrate does not improve oral glucose tolerance in patients with type 2 diabetes. Nutr Res 2015; 35:674-680.
- 67. Ashor AW, Chowdhury S, Oggioni C, Qadur O, Brandt K, Ishaq A, Mathers JC, Saretzki G, Siervo M. Inorganic nitrate supplementation in young and old obese adults does not affect acute glucose and insulin responses but lowers oxidative stress. J Nutr 2016; 146:2224-2232.
- 68. Gregory CM, Bickel CS. Recruitment patterns in human skeletal muscle during electrical stimulation. Phys Ther 2005;85:358-364.
- 69. Derave W, Taes Y. Beware of the pickle: health effects of nitrate intake. J Appl Physiol 2009;107:1677; author reply 1678.
- 70. Hord NG, Tang Y, Bryan NS. Food sources of nitrates and nitrites: the physiologic context for potential health benefits. Am J Clin Nutr 2009;90:1-10.
- 71. Kirby BS, Vovles WF, Simpson CB, Carlson RE, Schrage WG, Dinenno FA. Endothelium-derived vasodilation and exercise hyperemia in ageing humans: impact of acute ascorbic acid administration. J Physiol 2009;587:1989-2003.
- 72. Richards JC, Crecelius AR, Larson DG, Dinenno FA. Acute ascorbic acid ingestion increases skeletal muscle blood flow and oxygen consumption via local vasodilation during graded handgrip exercise in older adults. Am J Physiol Heart Circ Physiol 2015;309:H360-H368.
- 73. Buglioni A, Burnett JC Jr. New pharmacological strategies to increase cGMP. Ann Rev Med 2016;67:229-243.
- 74. Romero SA, Gagnon D, Adams AN, Moralez G, Kouda K, Jaffery MF, Cramer MN, Crandall CG. Folic acid ingestion improves skeletal muscle blood flow during graded handgrip and plantar flexion exercise in aged humans. Am J Physiol Heart Circ Physiol 2017;313:H658-H656.